CLINICAL TRIAL: NCT04429009
Title: A Randomized Control Trial of ZEPHYRx Gamified Incentive Spirometry Compared to Traditional Spirometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: My Music Machines Inc. (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZEPHYRx Rochester
Record Dates: First submitted 2020-05-12; First posted 2020-06-11 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Thoracic Surgery; Respiratory Therapy
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: All lobectomy and wedge resection patients meeting the inclusion criteria will be recruited (from the start of the study date until recruitment goal it reached) and consenting participants will be randomized to a study arm or a control arm. Each arm will consist of 50 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Study Group (Experimental): Participants in this group will be prescribed to use the ZEPHYRx RT device for incentive spectrometer once every hour during waking hours to perform a series of 10 deep breaths. The novel ZEPHYRx RT system consists three components:
  1. The Spirobank Smart Spirometer, which is a non-significant risk, FDA-cleared diagnostic spirometer made by Medical International Research (MIR) that connects via bluetooth to an Android tablet.
  2. A Samsung 10-inch tablet provided by Pad-in-Motion Inc. that will be connected to the hospital GuestWiFi network.
  3. The ZEPHYRx Respiratory Therapy video game application installed on the tablet. This application consists of seven games that have been created to combine traditional IS techniques with playing a breath controlled video game. The application will record data while playing the video games including date/time of use, game played, inhalation duration, and inhalation volume.
  Interventions: Device: ZEPHYRx Respiratory Therapy (RT) System
- Control Group (Active Comparator): Participants in this group will be prescribed to routine respiratory care, Routine respiratory care involves the use of a standard incentive spirometer that is not a digital device and does not include any built-in reminder. As per routine care, the nurse or respiratory therapist will remind the subjects to perform a series of at least 10 deep breaths every hour.
  Interventions: Device: Standard Incentive Spirometer

INTERVENTIONS:
Device: ZEPHYRx Respiratory Therapy (RT) System — A breath controlled video game system for respiratory therapy
  Arms: Active Study Group
Device: Standard Incentive Spirometer — A simple (not digital) plastic device that contains a piston that rises inside the device and measures the volume of your breath
  Arms: Control Group

SUMMARY:
The primary aim of this randomized control trial is to analyze by direct comparison the ZEPHYRx Respiratory Therapy (RT) system and the FDA approved standard of care (SOC) incentive spirometer (IS), used for FDA approved indications at the University of Rochester Medical Center (URMC). This comparison will determine subject preferences in terms of usability and simplicity of each, as well as subject engagement and adherence to the prescribed respiratory therapy routine. Additionally, the study will analyze the effectiveness of the gamified spirometry with regards to spirometry volumes, frequency of usage, and pulmonary complications 30 days post discharge.

DETAILED DESCRIPTION:
Lobectomy and wedge resection patients at University of Rochester Medical Center meeting the eligibility criteria will be screened and consented by members of the research team prior to surgery at their pre-operative clinic visit. Once a subject meets the inclusion criteria for this study, the subject will be randomly assigned to one of the two arms of this study by a flip of a coin. To ensure that we meet the predicted 50 subjects in each arm of the study, every second subject enrolled will be assigned to the opposite arm of the previously assigned subject.

Subjects enrolled in the study arm:

Following surgery or extubation, and once no longer under the influence of anesthesia, the patient enrolled into the study arm will be provided with a ZEPHYRx incentive spirometer device connected to an Amazon Kindle Fire HD Tablet. A respiratory therapist, nurse, doctor, or research team member will teach the subject how to use the device and the tablet, and walk them through the first series of breaths. A built-in bell reminder in the device will ring once every hour between the hours of 8:00 a.m. and 8:00 p.m. to remind patients to use the device, this feature is part of the research and a feature programmed into the device. Additionally, subjects will answer questions on their tablet about pain level on a scale of 0-10 before and after each round of game play. At discharge, the subjects in the study arm will return their assigned tablet and will be issued a standard incentive spirometer to continue respiratory therapy at home, per standard of care. Subjects in the study arm will not be held responsible for lost, stolen or damaged tablets or incentive spirometers. The subject in the study arm may choose to keep or discard the ZEPHYRx incentive spirometer device. The device will record subject usage, including number of breaths, number of sessions, total time the device was in use, inspiratory volumes, and pain level (0-10) before and after each round of game play.

Subjects enrolled in the control arm:

Following surgery or extubation, and once no longer under the influence of anesthesia, the patient enrolled in the control arm will meet with an RT, nurse, doctor, or research team member to receive an FDA approved incentive spirometry device and appropriate training thus initiating the study. Routine respiratory care involves the use of a standard incentive spirometer that is not a digital device and does not include any built-in reminder. As per routine care, the nurse or respiratory therapist will remind the subjects in both arms of the study to perform their respiratory therapy of at least 10 breaths per hour. In order to obtain data comparable to what the ZEPHYRx respiratory therapy system will collect, similar data will be collected from subjects in the control arm on a data sheet by an RT, nurse, doctor, or research team member 3 times a day until the subject is discharged. The only questionnaire will be the standard of care pain scale questions which the subjects in the control arm will have to complete in written form. Upon discharge, subjects in the control arm of the study will be allowed to keep their standard of care incentive spirometer in order to continue respiratory therapy at home, per standard of care. Subjects in the control arm will not be held responsible for lost, stolen or damaged incentive spirometers.

On a daily basis, a member of the research team will check that the device(s) is/are working correctly and will answer any questions the subject may have regarding the study or device.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients ages 18+ undergoing thoracic lobectomy surgery or wedge resection for tumor/nodule excisionat the University of Rochester Medical Center.

Exclusion Criteria:

* Patients under the age of 18
* Patients with diminished physical or mental capacity that make them incapable of operating a standard spirometer device
* Patients with visual or hearing impairments that make it difficult to understand verbal or written instructions
* Patients who are not able to read the language the ZEPHYRx software is available in (currently available only in English)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to prescribed spirometry routine | From extubation post-surgery to hospital discharge (estimated average of 2-4 days)
  Number of deep breaths taken per day with the prescribed device
Lung Volume | From extubation post-surgery to hospital discharge (estimated average of 2-4 days)
  Average daily inspiratory volume of the breaths taken with the prescribed device. Recorded 3 times per day by nurse or RT for the control group, and recorded at each use by the device for the active study group
Hospital Readmission | 30 days post discharge
  Hospital Readmission within 30 days of discharge

SECONDARY OUTCOMES:
Atelectasis | Evaluated for any required x-ray procedures during length of post-operated hospital stay (estimated 2-4 days per patient)
  Degree of Atelectasis assessed from chest radiography on a 5 point scale, where high scores correspond to more severe disease (1. no apparent disease, 2. subsegmental atelectasis, 3. segmental atelectasis, 4. lobar atelectasis, or 5. pneumonia)
Device Usability | At time of discharge (estimated to be 2-4 days post surgery extubation)
  A brief survey including likert scale questions on usability, and open ended feedback. Questions will be asked on a 5 point scale (1. strongly agree, 2. somewhat agree, 3. Neutral, 4. somewhat disagree, strongly disagree), with lower scores corresponding to better acceptance of the device.
Pain Scale pre and post exercises | Recorded before and after each session with the device for the treatment group, and by a nurse via paper survey 3 times per day for the control group during the length of hospital stay (estimated 2-4 days per patient)
  A measure of pain on the 0-10 Wong-Baker FACES pain scale that uses images of faces to determine pain level. 0 = no hurt (happy face), 10 = worst hurt (crying face)
Length of Stay | From extubation post-surgery to hospital discharge (estimated average of 2-4 days)
  Post Operative Hospital Length of Stay

CONTACTS AND LOCATIONS:
Overall Officials: Michal Lada, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No